CLINICAL TRIAL: NCT03385369
Title: A Phase 1, Randomized, Blinded, Single Ascending Dose Study to Evaluate the Safety and Pharmacokinetics of MEDI0382 in Overweight/Obese Subjects of Japanese or Chinese Descent
Brief Title: A Study to Evaluate the Safety and Pharmacokinetics of MEDI0382 in Overweight/Obese Subjects of Japanese or Chinese Descent
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: D5670C00012
Record Dates: First submitted 2017-11-29; First posted 2017-12-28 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Safety; Healthy Subjects
Keywords: MEDI0382; Safety; Tolerability; Pharmacokinetics; Immunogenicity
MeSH Terms: interventions — cotadutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Placebo Japanese Descent (Placebo Comparator): Participants of Japanese descent will receive a single subcutaneous injection of placebo matching to MEDI0382.
  Interventions: Drug: Placebo
- MEDI0382 50 mcg Japanese Descent (Experimental): Participants of Japanese descent will receive a single subcutaneous dose of 50 mcg MEDI0382.
  Interventions: Drug: MEDI0382
- MEDI0382 100 mcg Japanese Descent (Experimental): Participants of Japanese descent will receive a single subcutaneous dose of 100 mcg MEDI0382.
  Interventions: Drug: MEDI0382
- MEDI0382 150 mcg Japanese Descent (Experimental): Participants of Japanese descent will receive a single subcutaneous dose of 150 mcg MEDI0382.
  Interventions: Drug: MEDI0382
- Placebo Chinese Descent (Experimental): Participants of Chinese descent will receive a single subcutaneous injection of placebo matching to MEDI0382.
  Interventions: Drug: Placebo
- MEDI0382 100 mcg Chinese Descent (Experimental): Participants of Chinese descent will receive a single subcutaneous dose of 100 mcg MEDI0382.
  Interventions: Drug: MEDI0382

INTERVENTIONS:
Drug: MEDI0382 — Single dose of MEDI0382
  Arms: MEDI0382 100 mcg Chinese Descent; MEDI0382 100 mcg Japanese Descent; MEDI0382 150 mcg Japanese Descent; MEDI0382 50 mcg Japanese Descent
Drug: Placebo — Single dose of placebo
  Arms: Placebo Chinese Descent; Placebo Japanese Descent

SUMMARY:
This is a phase I, randomized, blinded study to evaluate the safety and pharmacokinetics of MEDI0382 following single dose administration to overweight/obese subjects of Japanese or Chinese descent

DETAILED DESCRIPTION:
This is a phase I, randomized, blinded study to evaluate the safety, tolerability, pharmacokinetics and immunogenicity of MEDI0382 following single dose administration to overweight/obese but otherwise healthy adult male and female subjects of Japanese or Chinese descent

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria:

1. Healthy subjects age 18 to 65 years inclusive at the time of consent.
2. Written informed consent and any locally required authorization (eg, Health Insurance Portability and Accountability Act in the USA), obtained from the subject prior to performing any protocol-related procedures, including screening evaluations.
3. Female subjects of childbearing potential must have a negative serum or urine pregnancy test at screening and randomization, and must not be lactating.
4. Females of childbearing potential who are sexually active with a nonsterilized male partner must use at least one highly effective method of contraception from screening and must agree to continue using such precautions through to the end of the study. It is strongly recommended for the male partner of a female subject to also use male condom plus spermicide throughout this period. Cessation of contraception after this point should be discussed with a responsible physician. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception.
5. Subject has a body weight ≥ 50 kg (110 lbs) and a BMI ≥ 23 and ≤ 40 kg/m2 inclusive.
6. Venous access suitable for multiple cannulations.

   Part A only:
7. Subject is a native of Japan or a Japanese American; defined as having both parents and four grandparents who are Japanese. This includes second and third generation subjects of Japanese descent whose parents or grandparents are living in a country other than Japan.

Part B only:

8. Subject is a native of China or a Chinese American; defined as having both parents and four grandparents who are Chinese. This includes second and third generation subjects of Chinese descent whose parents or grandparents are living in a country other than China.

____________________________________________________________

Exclusion Criteria:

Any of the following would exclude the subject from participation in the study:

1. Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results. Specific examples are:

   1. Past history of acute or chronic pancreatitis, or pancreatic amylase or lipase greater than twice the upper limit of normal (ULN) at screening.
   2. Past history of gastroparesis requiring treatment.
   3. Past history of surgery affecting the upper GI tract likely to affect the interpretation of safety and tolerability data.
   4. History of cholelithiasis leading to episodes of acute cholecystitis not treated by cholecystectomy, or known biliary disease.
   5. History of or family history of multiple endocrine neoplasia type 2; or serum calcitonin suggestive of thyroid C-cell hyperplasia (calcitonin level > 50 ng/L); or medullary thyroid carcinoma at screening.
   6. Past history of clinically significant cardiac rhythm disturbance (eg, permanent or paroxysmal atrial fibrillation/flutter, paroxysmal supraventricular tachycardia, paroxysmal ventricular tachycardia, presence of an implantable pacemaker device or cardioverter/defibrillator).
   7. History of treated or symptomatic cardiac failure.
   8. Impaired renal function, defined as estimated glomerular filtration rate < 60 mL/minute/1.73 m2 at screening.
2. History of previous myocardial infarction or cerebrovascular accident (eg, stroke).
3. History or presence of GI, renal, or hepatic disease (with the exception of Gilbert's syndrome), or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
4. History of cancer, with the exception of non-melanoma skin cancer.
5. Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks prior to dosing.
6. Positive hepatitis B surface antigen or hepatitis C virus antibody serology at screening.
7. Positive human immunodeficiency virus test at screening or use of antiretroviral medications as determined by medical history or subject's verbal report.
8. Any of the following based on screening blood tests:

   1. Aspartate aminotransferase (AST) ≥ 1.5 × ULN.
   2. Alanine aminotransferase (ALT) ≥ 1.5 × ULN.
   3. Total bilirubin ≥ 1.5 × ULN.
   4. Hemoglobin below 12 g/dL.
   5. Neutrophils < 1.5 × 10^9/L.
   6. Thyroid stimulating hormone level above the normal range.
9. Use of any of the following medicinal products:

   1. Concurrent or previous use of a GLP-1 receptor agonist.
   2. Current or previous use of systemic corticosteroids within the past 28 days prior to screening.
   3. Use of any licensed medicinal products, or herbal preparations for control of body weight or appetite, is prohibited from one week prior to Day -1 through Day 3.
10. Abnormal vital signs after 10 minutes of supine rest, defined as any of the following:

    1. Systolic BP < 90 mmHg or ≥ 140 mmHg.
    2. Diastolic BP < 50 mmHg or ≥ 90 mmHg.
    3. Heart rate < 45 or > 85 beats per minute.
11. Any clinically important abnormalities in rhythm, conduction (eg, Wolff-Parkinson-White syndrome, sick-sinus syndrome), or morphology of the resting 12-lead ECG, or any abnormalities in the ECG that, in the opinion of the investigator, may interfere with the interpretation of changes in the QTc, including abnormal T-wave morphology, or left ventricular hypertrophy.
12. Prolonged QTc using the Fridericia formula (QTcF) > 450 milliseconds, or shortened QTcF < 340 milliseconds based on 12-lead ECG, or family history of long QT syndrome.
13. PR (PQ) interval shortening < 120 milliseconds (PR < 120 but > 110 milliseconds is acceptable if there is no evidence of ventricular pre excitation).
14. PR (PQ) interval prolongation (> 240 milliseconds), intermittent second degree block (Wenckebach block while asleep is not exclusive) or third degree block, or atrioventricular dissociation.
15. Complete or intermittent complete bundle branch block, incomplete bundle branch block,or intraventricular conduction delay with QRS > 110 milliseconds. Subjects with QRS > 110 but < 115 milliseconds are acceptable if there is no evidence of ventricular hypertrophy.
16. Known or suspected history of drug abuse within the past 3 years as judged by the investigator.
17. History of alcohol abuse or excessive intake of alcohol within the past 3 years as judged by the investigator.
18. Positive screen for drugs of abuse or positive breath test for alcohol at screening. Subjects who use benzodiazepines for chronic anxiety or sleep disorders may be permitted to enter the study.
19. History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity as judged by the investigator.
20. Whole blood or red blood cell donation, or any blood loss > 500 mL within 2 months prior to screening.
21. Receipt of another new chemical entity (defined as a compound that has not been approved for marketing), or participation in any other clinical study that included drug treatment within at least 30 days or 5 half-lives of the administration of investigational product in this study (whichever is longer). The period of exclusion will end 30 days or 5 half-lives of investigational product after the final dose, whichever is longest. Subjects consented and screened, but not randomized into this study or a previous study, will not be excluded.
22. Psychiatric illness such that subjects have been committed to an institution by way of official or judicial order.
23. The subject is an employee, or close relative of an employee, of AstraZeneca, MedImmune, the CRO, or the study site, regardless of the employee's role.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2018-04-12 (Actual); Study Completion 2018-04-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs) | Day 1 through Day 29
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug and up to Day 29.
Number of Participants With Treatment Emergent Adverse Events of Special Interest (AESIs) | Day 1 through Day 29
  An AESI (serious or non-serious) was one of scientific and medical interest specific to understanding of study drug and may have required close monitoring and rapid communication by investigator to the sponsor.
Number of Participants With Abnormal Electrocardiogram (ECG) Reported as TEAEs | Day 1 through Day 29
  Number of participants with TEAEs related to clinically significant ECG abnormalities are reported.
Number of Participants With Vital Signs Abnormalities Reported as TEAEs | Day 1 through Day 29
  Number of participants with TEAEs related to vital sign abnormalities are reported.
Number of Participants With Abnormal Laboratory parameters Reported as TEAEs | Day 1 through Day 29
  Number of participants with TEAEs related to clinically significant abnormal laboratory parameter are reported.

SECONDARY OUTCOMES:
Number of Participants With Postive Anti-Drug Antibodies (ADA) Titer to MEDI0382 | Baseline (Day-1), Day 8, and Day 29
  The number of participants with positive serum antibodies to MEDI0382 are reported.
Maximum Observed Plasma Concentration (Cmax) of MEDI0382 | Pre dose; and at 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours post dose
Area Under the Concentration-time Curve From Time Zero to Infinity (AUC0-inf) of MEDI0382 | Pre dose; and at 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours post dose
Area Under the Concentration-time Curve From Time Zero to Last Time of Quantifiable Concentration (AUC0 last) of MEDI0382 | Pre dose; and at 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours post dose
Time to Maximum Observed Plasma Concentration (tmax) of MEDI0382 | Pre dose; and at 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours post dose
Apparent Terminal Elimination Half-life (t1/2) of MEDI0382 | Pre dose; and at 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours post dose
Apparent Clearance (CL/F) of MEDI0382 | Pre dose; and at 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Winkle, MD, FACP, FACG, CPI, Principal Investigator — Anaheim Clinical Trials LLC
Locations (1):
- Research Site, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: Undecided